CLINICAL TRIAL: NCT01861548
Title: Polish Mother and Child Cohort Study (REPRO_PL).Follow up of the Children.
Brief Title: Polish Mother and Child Cohort Study (REPRO_PL) - Follow up of the Children.
Acronym: REPRO_PL
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Prof., Medical University of Lodz
Other Study IDs: PBZ-MEiN-/8/2//2006; PNRF-218-AI-1/07 (Other Grant/Funding Number: Norwegian Financial Mechanism)
Record Dates: First submitted 2013-05-17; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Asthma; Atopic Dermatitis; Food Allergy; Wheezing
MeSH Terms: conditions — Asthma; Dermatitis, Atopic; Food Hypersensitivity; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, hair, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children (up to 24 months after birth): Investigators include into the study children delivered from women observed starting from between 8-12 weeks of single pregnancy, not assisted with reproductive technology, and not expected to be finished as spontaneous abor-tion. All women with the serious chronic diseases specified in study protocol such as diabetes, hypertension, nephrop-athy, epilepsy and cancer are excluded from the study. The same refers to suspicion of serious child malformations known to exist at the inclusion into the study.

SUMMARY:
The Polish Mother and Child Cohort is multicentre prospective study on different exposures.

Prospective cohort study design enables identification of exposures that may influence pregnancy outcome and chil-dren's health, verification of such exposures by biomarker measurements and notification of any changes in exposure levels.

The aim of the study is to evaluate the impact of exposure to different environmental factors during pregnancy and after birth on pregnancy outcome and children's health. Specific research hypotheses refer to the role of heavy metals, exposure to polycyclic aromatic hydrocar-bons (PAHs) and environmental tobacco smoke (ETS) in the aetiology of intrauterine growth retardation (IUGR), preterm delivery (PD) and the risk of respiratory diseases, allergy and poor mental and physical development. It is also intended to explain the role of oxidative stress and nutritional status of the pregnant women. The impact of occupational exposures and stressful situations on pregnancy outcome will be evaluated from question-naire data.

The results of the study will help to determine levels of child prenatal and postnatal exposure in several areas of Poland and their im-pact on course and outcome of pregnancy and children's health.

This protocol concerns the children that are followed-up from birth to the age of 2 years to determine long term effects of pre- and postnatal environmental exposures.

DETAILED DESCRIPTION:
The Polish Mother and Child Cohort is multicentre prospective study on different exposures.

Prospective cohort study design enables identification of exposures that may influence pregnancy outcome and chil-dren's health, verification of such exposures by biomarker measurements and notification of any changes in exposure levels.

The aim of the study is to evaluate the impact of exposure to different environmental factors during pregnancy and after birth on pregnancy outcome and children's health. Specific research hypotheses refer to the role of heavy metals, exposure to polycyclic aromatic hydrocar-bons (PAHs) and environmental tobacco smoke (ETS) in the aetiology of intrauterine growth retardation (IUGR), preterm delivery (PD) and the risk of respiratory diseases, allergy and poor mental and physical development. It is also intended to explain the role of oxidative stress and nutritional status of the pregnant women. The impact of occupational exposures and stressful situations on pregnancy outcome will be evaluated from question-naire data.

The results of the study will help to determine levels of child prenatal and postnatal exposure in several areas of Poland and their im-pact on course and outcome of pregnancy and children's health.

This protocol concerns the children that are followed-up from birth to the age of 2 years to deter-mine long term effects of pre- and postnatal environmental exposures.

Exposure of children to ETS. Postnatal children exposure to ETS at 12, and 24 months after birth is assessed. From the children urine sample and saliva samples from mothers who will declare smoking abstinence are collected. The saliva and urine cotinine level is analysed using high performance liquid chromatography coupled with tandem mass spectrometry/positive electrospray ionization (LC-ESI+MS/MS) and isotope dilution.

Exposure of children to PAH. The HPLC technique is used for the analysis of the level of 1-hydroksypyrene in urine as the biomarker of PAH exposure (12 and 24 months).

Exposure to lead, cadmium, mercury in children. Blood and hair are collected for about 100 children. Total and inorganic mercury is analyzed using cold vapour atomic fluorescence spectrophotometry. The lead and cadmium concentrations in blood is determined by graphite-furnance atomic-absorption spectrometry.

Exposure to indoor allergens, endotoxins and glucans. The analyzis is covered approx. 50 family homes of children. The settled dust is collected from floors in leaving rooms and in children beds (mattresses and blankets). To determine allergens concentrations in dust samples, the commercially available enzymelinked immunosorbent assey (ELISA) kits ispplied according to the protocol.To determine endotoxins and (1→3)-β-D-glucans concentrations the LAL test will be applied. The questionnaire study is performed among parents in order to obtain the data about demographic factors and home conditions.

Questionnaires conducted with mothers 12, and 24 months after delivery. Mothers of all children are interviewed. The questionnaires investigate the children's health and development, the nutrition of the small child and their contacts with other children. The smoking status of the parents and other potential sources of children's ETS exposure are identified. Information about proximity to heavy traffic is inquired. Additionally the information from the closets to his/her place of living air pollution monitoring station is collected. Exposure to other environmental factors including domestic animals, home dust, household cleaning agents and indoor used pesticides is evaluated by the questionnaire.

Determination of the prevalence of the upper and lower respiratory tract infections, middle ear diseases and allergy among the child. The incidence of the upper and lower respiratory tract infections, middle ear diseases and symptoms of allergy among the child is identified based on the detailed interview with the mothers in 12 and 24 month after child birth. This interviews is conducted by paediatricians. For each child upper and lower respiratory tract infections (tonsillitis, laryngitis, bronchitis and pneumonia), as well as middle ear diseases and allergy to food and inhalant allergens is identified based on the review of their medical charts. The duration of each infection and disease, medications taken and hospitalization is identified. The current health status of the chid and child' anthropometry (high, weight) is preformed by pediatrician.

Determination of the neurodevelopment of the children. BSID-III is used for assessment of child neurodevelopment. The tests is scheduled on 12 and/ 24 months of live and is conducted by psychologist or child development specialist. The test assesses five developmental areas of the child: cognitive, motor (fine and gross motor), language (receptive, expressive), social-emotional and adaptive behavior.

ELIGIBILITY:
Inclusion Criteria:

* Investigators include into the study children delivered from women observed starting from between 8-12 weeks of single pregnancy, not assisted with reproductive technology, and not expected to be finished as spontaneous abor-tion. All women with the serious chronic diseases specified in study protocol such as diabetes, hypertension, nephrop-athy, epilepsy and cancer are excluded from the study. The same refers to suspicion of serious child malformations known to exist at the inclusion into the study.

Exclusion Criteria:

* Serious child malformations known to exist at the inclusion into the study.
* Children delivered from all women with the serious chronic diseases specified in study protocol such as diabetes, hypertension, nephrop-athy, epilepsy and cancer are excluded from the study.

Ages: 1 Minute to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Investigators include into the study children delivered from women observed starting from between 8-12 weeks of single pregnancy, not assisted with reproductive technology, and not expected to be finished as spontaneous abor-tion. All women with the serious chronic diseases specified in study protocol such as diabetes, hypertension, nephrop-athy, epilepsy and cancer are excluded from the study. The same refers to suspicion of serious child malformations known to exist at the inclusion into the study.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2007-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Exposure of children to Environmental tobacco smoke(ETS) | Change from baseline of exposure of children to environmental tobacco smoke at 12 months
  Postnatal children exposure to ETS at 12, and 24 months after birth is assessed. From the children urine sample and saliva samples from mothers who will declare smoking abstinence are collected. The saliva and urine cotinine level is analysed using high performance liquid chromatography coupled with tandem mass spectrometry/positive electrospray ionization (LC-ESI+MS/MS) and isotope dilution.

SECONDARY OUTCOMES:
Exposure of children to polycyclic aromatic hydrocarbons (PAH) | Change from baseline of exposure of children to polycyclic aromatic hydrocarbons at 12 months
  The high performance liquid chromatography (HPLC) technique is used for the analysis of the level of 1-hydroksypyrene in urine as the biomarker of PAH exposure.
Exposure to lead, cadmium, mercury in children. | Change from baseline of exposure to lead, cadmium, mercury in children at 12 months.
  Blood and hair are collected for about 100 children. Total and inorganic mercury is analyzed using cold vapour atomic fluorescence spectrophotometry. The lead and cadmium concentrations in blood is determined by graphite-furnance atomic-absorption spectrometry.
Exposure to indoor allergens, endotoxins and glucans in children. | Change from baseline of exposure to indoor allergens, endotoxins and glucans in children at 12 months.
  The analyzis is covered approx. 50 family homes of children. The settled dust is collected from floors in leaving rooms and in children beds (mattresses and blankets). To determine allergens concentrations in dust samples, the commercially available enzymelinked immunosorbent assey (ELISA) kits ispplied according to the protocol.To determine endotoxins and (1→3)-β-D-glucans concentrations the LAL test will be applied. The questionnaire study is performed among parents in order to obtain the data about demographic factors and home conditions.
Questionnaires conducted with mothers. | Change from baseline of questionnaires scores at 12 months.
  Mothers of all children are interviewed. The questionnaires investigate the children's health and development, the nutrition of the small child and their contacts with other children. The smoking status of the parents and other potential sources of children's ETS exposure are identified. Information about proximity to heavy traffic is inquired. Additionally the information from the closets to his/her place of living air pollution monitoring station is collected. Exposure to other environmental factors including domestic animals, home dust, household cleaning agents and indoor used pesticides is evaluated by the questionnaire.
Determination of the prevalence of the upper and lower respiratory tract infections, middle ear diseases and allergy among the child. | Change from baseline of the prevalence of infections and allergies at 12 months
  The incidence of the upper and lower respiratory tract infections, middle ear diseases and symptoms of allergy among the child is identified based on the detailed interview with the mothers in 12 and 24 month after child birth. This interviews is conducted by paediatricians. For each child upper and lower respiratory tract infections (tonsillitis, laryngitis, bronchitis and pneumonia), as well as middle ear diseases and allergy to food and inhalant allergens is identified based on the review of their medical charts. The duration of each infection and disease, medications taken and hospitalization is identified. The current health status of the chid and child' anthropometry (high, weight) is preformed by pediatrician.
Determination of the neurodevelopment of the children. | Change from baseline of the neurodevelopment of the children at 12 months
  Bayley Scales of Infant Development (BSID-III) is used for assessment of child neurodevelopment. The tests is scheduled on 12 and/ 24 months of live and is conducted by psychologist or child development specialist. The test assesses five developmental areas of the child: cognitive, motor (fine and gross motor), language (receptive, expressive), social-emotional and adaptive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MD,PhD,Prof., Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland; Monika Kopka, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland; Wojciech Hanke, MD,PhD,Prof., Principal Investigator — Nofer Institute of Occupational Medicine, Department of Environmental Epidemiology; Kinga Polanska, MD, PhD, Principal Investigator — Nofer Institute of Occupational Medicine, Department of Environmental Epidemiology
Locations (2):
- Poland (2):
  - Nofer Institute of Occupational Medicine, Department of Environmental Epidemiology, Lodz
  - Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, Lodz, Poland, Lodz

REFERENCES:
- [Derived] Podlecka D, Jerzynska J, Sanad K, Polanska K, Bobrowska-Korzeniowska M, Stelmach I, Brzozowska A. Micronutrients and the Risk of Allergic Diseases in School Children. Int J Environ Res Public Health. 2022 Sep 26;19(19):12187. doi: 10.3390/ijerph191912187. PMID 36231487
- [Derived] Stelmach I, Bobrowska-Korzeniowska M, Smejda K, Majak P, Jerzynska J, Stelmach W, Polanska K, Sobala W, Krysicka J, Hanke W. Risk factors for the development of atopic dermatitis and early wheeze. Allergy Asthma Proc. 2014 Sep-Oct;35(5):382-9. doi: 10.2500/aap.2014.35.3786. PMID 25295805
- [Derived] Stelmach I, Grzelewski T, Bobrowska-Korzeniowska M, Kopka M, Majak P, Jerzynska J, Stelmach W, Polanska K, Sobala W, Gromadzinska J, Wasowicz W, Hanke W. The role of zinc, copper, plasma glutathione peroxidase enzyme, and vitamins in the development of allergic diseases in early childhood: The Polish mother and child cohort study. Allergy Asthma Proc. 2014 May-Jun;35(3):227-32. doi: 10.2500/aap.2014.35.3748. PMID 24801465